CLINICAL TRIAL: NCT03052504
Title: Prospective Versus Retrospective Study of Comorbidity and Complications in Relation to Radical Cystectomy and Nephrectomy
Brief Title: Prospective Versus Retrospective Complications in Radical Cystectomy and Nephrectomy
Status: Completed | Type: Observational
Sponsor: Jørgen Bjerggaard Jensen (Other)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: CSA-1
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Bladder Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cx prospective: Cystectomy patients followed with prospective registration of complications
  Interventions: Other: Registration of complications
- Cx retrospective: Cystectomy patients followed with retrospective registration of complications
- Nx prospective: Nephrectomy patients followed with prospective registration of complications
  Interventions: Other: Registration of complications
- Nx retrospective: Nephrectomy patients followed with retrospective registration of complications

INTERVENTIONS:
Other: Registration of complications — Prospective registration
  Groups: Cx prospective; Nx prospective

SUMMARY:
The study will examine which differences there are in comorbidity and complications collected retrospectively from medical records compared with data collected prospectively in two groups of patients undergoing either radical cystectomy or radical nephrectomy.

Hypothesis is that he prevalence of registered comorbidity and minor complications in patients who have undergone radical cystectomy or nephrectomy, will increase if the data collection is focused and prospective, compared with retrospectively collected data.

The study will be conducted as a single-blind randomized controlled trial. Patients included in the study will be randomized to either control or intervention in the ratio 1:1. There are two groups of patients: Patients admitted to radical cystectomy and patients admitted to radical nephrectomy, due to cancer.

DETAILED DESCRIPTION:
Background:

Today there are many different systems to classify co morbidity and complication of radical cystectomy and nephrectomy. Regarding complication, there is Clavien Dindo classifications System and The National Surgical Quality Improvement Program (NSQIP) while Charlson Comorbidity Index (CCI) and Eastern Cooperative Oncology Group (ECOG) performance scale classifies comorbidity. At the present time, there is not a system that takes both parameters into account, although it is of high clinical relevance to be able to figure out the significant and important patient parameters that can influence the outcome of a treatment modality. Such a system is in development, from cystectomy patients, in this study's project group. This is currently to be validated in two large patient cohorts from respectively Herlev Hospital and Memorial Sloan Kettering Cancer Center, New York, USA. Virtually all previous publications on comorbidity or complications after cancer surgery, including the aforementioned, is based on data retrospectively collected from medical records. Even prospectively maintained database are based predominantly on data from records written in the journal prospective, but then transferred retrospectively to the database. The problem is that data on comorbidities and complications are not collected with this registration method in mind. Especially in the definition of the individual complications this contains a significant source of error. In addition, most minor complications that do not require re-intervention or re-operation, are probably underreported. Involvement of lesser complications after discharge is rarely reported, unless they lead to readmission. This is probably one of the causes of an uneven distribution in the reporting of serious complications requiring re-operation when comparing surgical case series, while the number of minor complications (Clavien 1-2) are highly variable. Even a minor complication which does not cause a readmission, can have a major impact on a patient's quality of life and experience of the disease. In addition, the small complications are often preventable, if you have a knowledge of their cause and context with the intervention. Patients who are to undergo cystectomy, are predominantly elderly patients with a large tobacco consumption and high comorbidity. At the same time cystectomy is associated with the highest risk of complications (75%) in cancer surgery, followed by nephrectomy patients (20%). Kidney cancer, and especially bladder cancer has a high- 1- and 5-year survivalrate. The patients will likely live for many years with their complications and the potential impact on quality of life as a result.

Since current knowledge and previous publications on comorbidity and/or complications after cancer surgery often is build on retrospective collected data, it will be highly relevant to examine the extent to which the retrospectively collected data is accurate by comparing with prospectively collected data. By conducting this study, it can be assessed which kind of gathering gives the correct information on the complications of radical cancer surgery and if previous publications should be revalidated?

Aim of the study The study will examine which differences there are in comorbidity and complications collected retrospectively from medical records compared with data collected prospectively.

Hypothesis The prevalence of registered comorbidity and minor complications in patients who have undergone radical cystectomy or nephrectomy, will increase if the data collection is focused and prospective, compared with retrospectively collected data.

Design The study will be conducted as a single-blind randomized controlled trial, as this form of study eliminates unknown confounders and have a high validity. Patients included in the study will be randomized to either control or intervention in the ratio 1:1. There are two groups of patients: Patients admitted to radical cystectomy and patients admitted to radical nephrectomy, due to cancer.

Study procedure In the control groups data on comorbidity and complications are collected retrospectively from medical records 90 days after the end of treatment, based on clearly defined criteria for comorbidity and complications, and severity of these (Clavien gradation). In the intervention group the investigator must collect information on comorbidity, preoperative, in a systematic review with a questionnaire in cooperation with the patient. Details about complications is collected daily at bedside, at rounds, by the investigator. Additionally, the patient receives a questionnaire at discharge. This must be answered at home. The investigator and the patient will go through the questionnaire at the first visit to the ambulatory. A second and identical questionnaire, in a stamped envelope, is handed out to the patient. In the last two questionnaires the patient must record contact with the family doctor, emergency physician, nurse and other hospital departments. Furthermore, any kind of medicine, pain or disability must be described. In the intervention group the same defined criteria are used as in the control group. Physicians involved in the management of the patient, is blinded to the group to which the patient is randomly assigned to, and is thus unaware of whether the patient is in the intervention group or the control group. Subsequently for the intervention group a retrospective collection of data from medical records is made and compared with the control group. This ensures that the randomization has been sufficient.

Primary endpoints

* Prevalence of procedure related complications (Clavien score)

  * During hospitalization postoperative before discharge
  * Within the first week after discharge
  * Within the second week after discharge
* Prevalence of preoperative comorbidity

Secondary Endpoints

* Patient comorbidity: Acute myocardial infarction, angina pectoris, arrhythmias, previous cardiac surgery, venous diseases, hypertension, hypercholesterolemia, abdominal aortic aneurysm, claudicatio, chronic obstructive pulmonary disease, peptic ulcer, alcohol abuse, liver disease, stroke, diabetes mellitus type I and II, connective tissue disease, osteoporosis, kidney transplant, kidney failure, leukemia/lymphoma, previous malignant disease with & without metastases.
* Patient complication: antiemetics, antipyretics, antibiotics, diuretics, VAS (Visual Analog Pain Scale) score, newly started or increased help from home care, newly started or more visits from the home nurse, newly started physical therapy, blood transfusion
* Is there a significant variation in comorbidity collected from questionnaires and medical records, respectively.

Statistics and sample size The number of patients in the study is based on the following assumptions: For the cystectomy- and nephrectomy patients with complications retrospectively calculated, it is assumed that complications that needs intervention is detected respectively about 50% and 20%. This is in accordance with the highest indication in major international surveys with retrospective registering. Based on previous experiences, the real number is estimated to be respectively minimum 85% and 35%. With an alpha value at 0,05 and a beta value at 0,20, this gives a required number of patients at 66 for cystectomy patients and 90 nephrectomy patients, to be able to demonstrate a significant difference.

Statistical analyses will be performed with primarily non-parametric test using MedCalc for Windows, version 15.8 or later (MedCalc Software, Ostend, Belgium).

Data management Patients will be enrolled after signing informed consent. Patient data will be entered directly into the electronic CRF (Clinical Registration Form) on a secure server using REDCap, which is a secure server based system with a security that exceeds the demands and guidelines of "Persondataloven" and is recommended by Aarhus University. Data are stored according to regulations by the Danish Data Protections Agency.

Perspectivation If the study concludes that the project groups classification system is based on valid data and find out what kind of data collection that provides the most accurate picture of the patients relationship between co-morbidities and complications, we will in future be able to give patients more individualized treatment. This is desirable both for the patient and the therapist. In this way the study classification system will be able to avoid the patient living a life with post operative complications and a complicated treatment. This will also be able to reduce the use of health care resources, that can then be uses elsewhere.

Ethical considerations The study will be conducted in accordance with the protocol, applicable regulatory requirements and the ethical principles of the Declaration of Helsinki as adopted by the 18th World Medical Assembly in Helsinki, Finland in 1064 and subsequent versions.

The patients that by informed consent is included in the study, are exposed neither to different surgery or other treatment than they would have been without participation in the study. The extra interviews and daily rounds will attempt established in connection with the patient's usual attendance and stay at the hospital, to avoid extra visits. There must be calculated some extra time spent in connection with participation in the trial. Studies show that patients in scientific studies, feel that they receive a better treatment.

The study is approved in the Data Inspectorate and assessment is ongoing in the Research Ethics Committee, where approval is mandatory before starting.

Project feasibility The study is performed in an internationally acknowledged research environment at department of urology, Aarhus University Hospital, Skejby. Baseline data are collected until approximately May 2017 and follow-up data August 2017. This means that data will be available in time to complete the thesis and a paper for publication. The research year student will be affiliated to the department. All necessary analysis methods are established in the department, and hardware and software will be provided.

ELIGIBILITY:
Inclusion criteria

* Age > 18 years
* Competente and able individuals
* Consented participation
* Planned radical cystectomy or nephrectomy due to cancer Exclusion criteria
* Failure to consent to participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cystectomy or nephrectomy
Sampling Method: Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Severety of postoperative complications | 90 days
  Clavien grading

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No